CLINICAL TRIAL: NCT01704326
Title: A Prospective, Multicenter Consecutive Series Study of Patients Treated With the Journey Deuce Bicompartmental Knee System
Brief Title: A Study of Patients Treated With the Journey Deuce Bicompartmental Knee System
Status: Completed | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DEUK01
Record Dates: First submitted 2012-09-24; First posted 2012-10-11 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: Osteoarthritis
Keywords: Deuce; Journey Deuce; Knee pain; Osteoarthritis; Bicompartmental; Femoral; Medial
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a prospective, multicenter, consecutive clinical study of the Journey Deuce Knee System and is intended to evaluate the safety and effectiveness of the new device.

DETAILED DESCRIPTION:
The objectives of this study are to assess the safety and effectiveness of the Journey Deuce Bicompartmental Knee System. Patients will be examined clinically at time intervals throughout the study duration. Exams will include completion of clinical assessment, x-rays, and completion of patient questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Patient presents with non-inflammatory degenerative joint disease of the medial and patellofemoral compartments requiring a unilateral knee replacement.
* Patient is 30 to 75 years of age, inclusive.
* Patient is willing to consent to participate in the study by signing and dating an IRB-approved consent form.
* Patient plans to be available for follow-up through five years postoperative.

Exclusion Criteria:

* Patient is known to have insufficient femoral or tibial bone stock resulting from conditions such as cancer, distal femoral/proximal tibial osteotomy, significant osteoporosis or metabolic bone disorders.
* Patient is immunosuppressed, has an autoimmune disorder, or an immunosuppressive disorder (i.e. chronic condition characterized by markedly inhibited ability to respond to antigenic stimuli.) Examples of such conditions include patients who are on immunosuppressive therapy (corticosteroid hormones in large amounts, cytotoxic drugs, antilymphocytic serum or irradiation in large doses) or patients with acquired immunodeficiency syndrome (AIDS).
* Patient has inflammatory arthritis (e.g. rheumatoid arthritis)
* Patient has BMI greater than or equal to 40.
* Patient has had major knee surgery in the past i.e. HTO, unicondylar knee replacement, failed fracture fixation.
* Patient has an active infection, local or systemic.
* Patient has physical, emotional or neurological conditions that would compromise the patient's compliance with postoperative rehabilitation and followup (e.g.: drug or alcohol abuse, serious mental illness, or general neurological conditions such as Parkinson, Multiple sclerosis, etc.).
* Patient has ACL deficiency in the study knee.
* Patient has hip arthritis and/or replacement.
* Patient has lateral compartment disease.
* Patient is pregnant or plans to become pregnant during the course of the study.
* Patient has a known sensitivity to materials in the device.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients eligible for this study are non-inflammatory degenerative joint disease patients requiring a primary unilateral knee surgery. The affected areas must be limited to the medial and patellofemoral compartments.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2006-09; Primary Completion 2012-02 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Change in Knee Society Score | Preoperative-2 years
  Assess knee pain, function and range of motion using the Knee Society Clinical Rating System

SECONDARY OUTCOMES:
Oxford Knee Outcome Questionnaire | Preoperative, 6 weeks, 3 months, 6 months, 1 year and 2 years
  Patient evaluation of function
Radiographic Evaluation | 6 weeks, 1 year and 2 years
  X-rays will be assessed for evidence of implant loosening, surface wear, migration or any other clinical or radiographic abnormalities.
Patient Satisfaction | 6 weeks, 3 months, 6 months, 1 year and 2 years
  Patient satisfaction questionnaire to be completed at each follow-up visit
Adverse Events | When Necessary
  All intra-operative, discharge, and post-operative surgical/hospitalization or study knee-related adverse events will be captured during the study to assess for safety issues.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Orthopaedic Center of Vero Beach, Vero Beach, Florida
  - Orthopaedic Surgery Specialists, Ltd., Park Ridge, Illinois
  - Henry County Center for Orthopedic Surgery & Sports Medicine, New Castle, Indiana
  - Iowa Orthopaedic Center, PC, Des Moines, Iowa